CLINICAL TRIAL: NCT07060287
Title: Predictive Value of miR-21 and miR-486 Expression in Patients Undergoing Clock-Guided Minimally Invasive Surgery for Pulmonary Nodules
Brief Title: Prognostic Value of miR-21 and miR-486 in Pulmonary Nodule Surgery
Status: Completed | Type: Observational
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yingchun Ren, Principal investigator, The First Hospital of Hebei Medical University
Other Study IDs: 2019S00479
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Nodule Cm
Keywords: miR-21; miR-486; clock-guided anatomical positioning; pulmonary nodules; survival analysis; VATS
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Intraoperatively resected pulmonary nodule tissues were collected, and total RNA was extracted for miRNA quantification.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High miR-21/miR-486 Expression Group (n=62): Patients whose resected pulmonary nodule tissue showed expression of miR-21 greater than a 2.5-fold change or miR-486 greater than a 1.8-fold change compared to reference levels, as determined by ROC curve analysis.
  Interventions: Procedure: Clock-Guided Minimally Invasive Surgery
- Low miR-21/miR-486 Expression Group (n=76): Patients whose resected pulmonary nodule tissue showed expression of miR-21 less than or equal to a 2.5-fold change and miR-486 less than or equal to a 1.8-fold change compared to reference levels.
  Interventions: Procedure: Clock-Guided Minimally Invasive Surgery

INTERVENTIONS:
Procedure: Clock-Guided Minimally Invasive Surgery — All participants underwent video-assisted thoracoscopic surgery (VATS) for pulmonary nodule resection. Nodule localization was performed using a clock-guided anatomical positioning technique with a 3D reconstruction system. The surgical procedure included wedge resection, segmentectomy, or lobectomy based on clinical judgment.

SUMMARY:
This study prospectively evaluated the prognostic value of microRNA-21 (miR-21) and microRNA-486 (miR-486) expression in patients with pulmonary nodules who underwent clock-guided minimally invasive surgery. The study aimed to determine if high expression levels of these miRNAs in resected nodule tissue correlate with poorer clinical outcomes, including larger residual tumor size, higher metabolic activity, and shorter overall and progression-free survival.

DETAILED DESCRIPTION:
Pulmonary nodules pose a significant diagnostic and therapeutic challenge. Clock-guided anatomical positioning is a novel technique that improves the precision of minimally invasive surgical resection. MicroRNAs, such as miR-21 and miR-486, are known to be involved in tumorigenesis and have been identified as potential biomarkers. This study was a prospective cohort study designed to investigate the prognostic significance of miR-21 and miR-486 expression in the context of this advanced surgical technique. A total of 138 patients undergoing clock-guided minimally invasive surgery for pulmonary nodules were enrolled. Intraoperative nodule tissues were collected to quantify miRNA expression levels via real-time PCR. Patients were then stratified into high-expression and low-expression groups based on predetermined cut-off values. Postoperative outcomes, including residual nodule characteristics (size, density, metabolic activity) and survival data (Overall Survival and Progression-Free Survival), were collected and compared between the two groups to assess the predictive power of these miRNAs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Single or multiple pulmonary nodules confirmed by imaging;
* Pathologically confirmed or highly suspected malignancy;
* Eligible for clock-guided minimally invasive surgery;
* No contraindications to surgery;
* Signed informed consent.

Exclusion Criteria:

* Uncontrolled comorbidities (e.g., hypertension >180/110 mmHg, HbA1c >9%);
* Inoperable status;
* Benign nodules confirmed by pathology;
* Severe organ dysfunction (e.g., LVEF <40%, eGFR <30 mL/min);
* Immunosuppressive therapy;
* Recent anticancer treatment (<3 months);
* Lost to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprised 138 adult patients (age ≥18 years) with pulmonary nodules who were scheduled for clock-guided minimally invasive surgery at the Department of Thoracic Surgery, the First Hospital of Hebei Medical University. Participants were prospectively and consecutively enrolled if they had pathologically confirmed or highly suspected malignant nodules and met all predefined inclusion and exclusion criteria. All participants provided written informed consent prior to enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Assessed up to January 2022 (up to 24 months of follow-up)
  Defined as the time from the date of surgery to the date of death from any cause.
Progression-Free Survival (PFS) | Assessed up to January 2022 (up to 24 months of follow-up)
  Defined as the time from the date of surgery to the date of disease progression (local recurrence or distant metastasis) or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Residual Nodule Size | Assessed at 6 months postoperatively
  Measurement of the maximum diameter (in cm) of any residual or recurrent nodule on chest CT scans.
Residual Nodule Density | Assessed at 6 months postoperatively
  Measurement of the density of any residual or recurrent nodule in Hounsfield Units (HU) on non-contrast chest CT scans.
Residual Nodule Metabolic Activity | Assessed at 6 months postoperatively
  Quantification of metabolic activity of any residual or recurrent nodule using the maximum standardized uptake value (SUVmax) on 18F-FDG PET/CT scans.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China